CLINICAL TRIAL: NCT03170349
Title: The CLASP Study Edwards PASCAL TrAnScatheter Mitral Valve RePair System Study
Acronym: CLASP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-05
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Results first posted 2021-12-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Mitral Valve Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Edwards PASCAL Transcatheter Mitral Valve Repair System (Experimental)
  Interventions: Device: Mitral Valve Repair

INTERVENTIONS:
Device: Mitral Valve Repair — Minimal Invasive Transcatheter Mitral Valve Repair

SUMMARY:
The purpose of this study is to assess the safety, performance and clinical outcomes of the Edwards PASCAL Transcatheter Mitral Valve Repair (TMVr) System.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety, performance and clinical outcomes of the Edwards PASCAL Transcatheter Mitral Valve Repair (TMVr) System. This is a multi-center, multi-national, prospective, single arm, safety, performance and clinical outcomes study.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated IRB/ethics committee approved study consent form prior to study related procedures
* Eighteen (18) years of age or older
* New York Heart Association (NYHA) Functional Class II-IVa heart failure despite optimal medical therapy
* Candidacy for surgical mitral valve repair or replacement determined by Heart Team evaluation
* Clinically significant mitral regurgitation (moderate-to-severe or severe mitral regurgitation) confirmed by transesophageal echocardiography (TEE) and transthoracic echocardiography (TTE).
* The primary regurgitant jet is non-commissural. If a secondary jet exists, it must be considered clinically insignificant.
* Mitral valve area (MVA) ≥ 4.0 cm² as measured by planimetry. If MVA by planimetry is not measurable, pressure half-time measurement is acceptable.

Exclusion Criteria:

* Patient in whom a TEE is contraindicated or screening TEE is unsuccessful
* Leaflet anatomy which may preclude PASCAL device implantation, proper device positioning on the leaflets, or sufficient reduction in mitral regurgitation.
* Mitral valve area (MVA) < 4.0 cm² as measured by planimetry (If MVA by planimetry is not measurable, PHT measurement is acceptable)
* Echocardiographic evidence of intracardiac mass, thrombus, or vegetation
* Physical evidence of right sided congestive heart failure and echocardiographic evidence of severe right ventricular dysfunction
* Concurrent medical condition with a life expectancy of less than 12 months in the judgment of the Investigator
* Patient is currently participating or has participated in another investigational drug or device clinical study where the primary study endpoint was not reached at time of enrollment
* Patient is under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2025-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gideon Cohen, MD, Principal Investigator — Sunnybrook Hospital; Ulrich Schafer, MD, Principal Investigator — BundeswehrZentralkrankenhaus Koblenz; Molly Szerlip, MD, Principal Investigator — The Heart Hospital Baylor
Locations (17):
- United States (8):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Colorado Denver, Aurora, Colorado
  - NorthShore University HealthSystem, Evanston, Illinois
  - Henry Ford Hospital, Detroit, Michigan
  - Morristown Medical Center, Morristown, New Jersey
  - Carolinas Medical Center, Charlotte, North Carolina
  - The Heart Hospital Baylor Plano, Plano, Texas
  - University of Virginia Health System, Charlottesville, Virginia
- Australia (2):
  - Metro North Hospital & Health Service, The Prince Charles Hospital, Brisbane, Chermside
  - Sydney Local Health District, Royal Prince Alfred Hospital, Camperdown, New South Wales
- Canada (3):
  - St. Paul's Hospital, Providence Health Care Research Institute, Vancouver, British Columbia
  - Sunnybrook Hospital, Toronto, Ontario
  - St Michael Hospital, Toronto, Ontario
- Universitaetsklinikum Bonn, Medizinische Klinik II, Kardiologie, Bonn, Germany
- Hygeia Hospital, Athens, Greece
- San Rafaelle Hospital, Milan, Italy
- Inselspital, University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Webb JG, Hensey M, Szerlip M, Schafer U, Cohen GN, Kar S, Makkar R, Kipperman RM, Spargias K, O'Neill WW, Ng MKC, Fam NP, Rinaldi MJ, Smith RL, Walters DL, Raffel CO, Levisay J, Latib A, Montorfano M, Marcoff L, Shrivastava M, Boone R, Gilmore S, Feldman TE, Lim DS. 1-Year Outcomes for Transcatheter Repair in Patients With Mitral Regurgitation From the CLASP Study. JACC Cardiovasc Interv. 2020 Oct 26;13(20):2344-2357. doi: 10.1016/j.jcin.2020.06.019. PMID 33092709
- [Derived] Lim DS, Kar S, Spargias K, Kipperman RM, O'Neill WW, Ng MKC, Fam NP, Walters DL, Webb JG, Smith RL, Rinaldi MJ, Latib A, Cohen GN, Schafer U, Marcoff L, Vandrangi P, Verta P, Feldman TE. Transcatheter Valve Repair for Patients With Mitral Regurgitation: 30-Day Results of the CLASP Study. JACC Cardiovasc Interv. 2019 Jul 22;12(14):1369-1378. doi: 10.1016/j.jcin.2019.04.034. Epub 2019 Jun 26. PMID 31255562

RESULTS

PARTICIPANT FLOW:
Groups:
- Edwards PASCAL Transcatheter Mitral Valve Repair System: Mitral valve repair with PASCAL implanted via transcatheter procedure
Period: At 30 Days Follow-up (±7 Days Window)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Started | 124
Completed | 123
Not Completed | 1
Not completed — Death | 1
Period: At 6 Months Follow-up (±30 Days Window)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Started | 123
Completed | 114
Not Completed | 9
Not completed — Death | 3
Not completed — Withdrawal by Subject | 1
Not completed — Exited for Other Reasons | 5
Period: At 1 Year Follow-up (±45 Days Window)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Started | 114
Completed | 106
Not Completed | 8
Not completed — Death | 6
Not completed — Exited for Other Reasons | 2
Period: At 2 Year Follow-up (±45 Days Window)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Started | 106
Completed | 88
Not Completed | 18
Not completed — Death | 13
Not completed — Withdrawal by Subject | 1
Not completed — Missed Visit | 4
Period: At 3 Year Follow-up (±45 Days Window)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Started | 92
Completed | 76
Not Completed | 16
Not completed — Death | 10
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2
Not completed — Missed Visit | 2
Period: At 4-year Follow-up (±45 Days Window)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Started | 78
Completed | 61
Not Completed | 17
Not completed — Death | 13
Not completed — Missed Visit | 2
Not completed — Exited for Other Reasons | 2

BASELINE CHARACTERISTICS:
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 69
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: inches] | 66.7 (4.1)
Weight [Mean (Standard Deviation); unit: pounds] | 165.4 (34.0)
Body Mass Index [Mean (Standard Deviation); unit: kilogram/meter square] | 26.2 (4.9)
Tobacco Use [Count of Participants; unit: Participants]
  Current daily smoker | 4
  Former daily smoker | 63
  Never | 57
EuroSCORE II [Mean (Standard Deviation); unit: Units on a scale] — The European System for Cardiac Operative Risk Evaluation (EuroSCORE) II is a risk model which allows the calculation of the risk of death after a heart operation. The higher the score, the higher the risk of an adverse outcome EuroScore II risk levels are as follows: Low risk: <8 Moderate risk: 8-10 High risk: >10 Population: Data unavailable for 8 patients.
  Units on a scale
    number analyzed (Participants) | 116
    (all) | 5.8 (5.4)
STS Mortality Score [Mean (Standard Deviation); unit: Units on a scale] — The STS score is a validated risk-prediction model for open surgery based on data from the STS National Adult Cardiac Surgery Database. In general, an STS predicted risk of surgical mortality of 4%-8% is considered intermediate risk and 8% or greater is considered high risk. As of November 15, 2018, The Society of Thoracic Surgeons released an updated short-term risk calculator to reflect the latest 2018 adult cardiac surgery risk models. The STS Calculator allows you to calculate a patient's risk of mortality and morbidities for the most commonly performed cardiac surgeries.
  Units on a scale | 4.6 (3.3)
NYHA Class [Count of Participants; unit: Participants] — NYHA Classification - The stages of heart failure: 1. Class I - No symptoms and no limitation in ordinary physical activity. 2. Class II - Mild symptoms and slight limitation during ordinary activity. 3. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest. 4. Class IV - Severe limitations. Experiences symptoms even while at rest. Population: Data unavailable for 1 patient.
  Participants
    Class I: number analyzed (Participants) | 123
    Class I | 0
    Class II: number analyzed (Participants) | 123
    Class II | 49
    Class III: number analyzed (Participants) | 123
    Class III | 68
    Class IV: number analyzed (Participants) | 123
    Class IV | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Adverse Events (MAE)
Description: Composite of major adverse events (MAE) defined as cardiovascular mortality, stroke, myocardial infarction, new need for renal replacement therapy, severe bleeding and re-intervention for study device related complications at 30 days post-implant. MAEs during the first year of post-implant follow-up were adjudicated by a Clinical Events Committee of independent heart specialist physicians.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 124
Participants | 10

2. Primary Outcome: Device Success
Description: Device is deployed as intended and the delivery system is successfully retrieved as intended at the time of the patient's exit from the cardiac catheterization laboratory.
Time Frame: Exit from the cardiac catheterization laboratory
Population: Per device analysis
Measure: Count of Units; unit: Device
Units Other Than Participants: Device
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 124
Number analyzed (Device) | 189
Device | 175

3. Primary Outcome: Number of Participants With Procedural Success
Description: Device success with evidence of mitral regurgitation reduction to ≤ 2+ (mild-moderate) at discharge and without the need for a surgical or percutaneous intervention prior to hospital discharge. Mitral regurgitation was assessed by independent echocardiographic core laboratory review of transthoracic echocardiography (TTE) imaging.
Time Frame: through discharge
Population: Participants with procedural success data available after collection of all study data for the Discharge visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 122
Participants | 115

4. Primary Outcome: Clinical Success
Description: Procedural success with evidence of MR reduction to ≤ 2+ (mild-moderate) and without MAEs at 30 days. Mitral regurgitation was assessed by independent echocardiographic core laboratory review of transthoracic echocardiography (TTE) imaging.
Time Frame: 30 days
Population: Participants with clinical success data available after collection of all study data for the 30-Day visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 121
Participants | 105

5. Secondary Outcome: Mitral Regurgitation Reduction
Description: Mitral regurgitation (MR) severity at 30 days, 6 months, 1 year and annually thereafter. Mitral regurgitation reduction was assessed by independent echocardiographic core laboratory review of transthoracic echocardiography (TTE) imaging.
Time Frame: Baseline, 30 Days, 6 Months, 1 Year, 2 Years, 3 Years, 4 Years
Population: Participants with an MR severity assessment available after collection of all study data for the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 124
Participants
  Baseline: None/Trace (0+) | 0
  Baseline: Mild (1+) | 1
  Baseline: Mild-Moderate (2+) | 0
  Baseline: Moderate-Severe (3+) | 66
  Baseline: Severe (4+) | 57
  30 Days: number analyzed (Participants) | 117
  30 Days: None/Trace (0+) | 18
  30 Days: Mild (1+) | 72
  30 Days: Mild-Moderate (2+) | 23
  30 Days: Moderate-Severe (3+) | 2
  30 Days: Severe (4+) | 2
  6 Months: number analyzed (Participants) | 111
  6 Months: None/Trace (0+) | 17
  6 Months: Mild (1+) | 64
  6 Months: Mild-Moderate (2+) | 28
  6 Months: Moderate-Severe (3+) | 2
  6 Months: Severe (4+) | 0
  1 Year: number analyzed (Participants) | 92
  1 Year: None/Trace (0+) | 13
  1 Year: Mild (1+) | 57
  1 Year: Mild-Moderate (2+) | 22
  1 Year: Moderate-Severe (3+) | 0
  1 Year: Severe (4+) | 0
  2 Years: number analyzed (Participants) | 71
  2 Years: None/Trace (0+) | 11
  2 Years: Mild (1+) | 40
  2 Years: Mild-Moderate (2+) | 18
  2 Years: Moderate-Severe (3+) | 2
  2 Years: Severe (4+) | 0
  3 Years: number analyzed (Participants) | 59
  3 Years: None/Trace (0+) | 10
  3 Years: Mild (1+) | 32
  3 Years: Mild-Moderate (2+) | 14
  3 Years: Moderate-Severe (3+) | 3
  3 Years: Severe (4+) | 0
  4 Years: number analyzed (Participants) | 45
  4 Years: None/Trace (0+) | 9
  4 Years: Mild (1+) | 28
  4 Years: Mild-Moderate (2+) | 5
  4 Years: Moderate-Severe (3+) | 2
  4 Years: Severe (4+) | 1

6. Secondary Outcome: All-cause Mortality
Description: All-cause mortality at 30 days, 6 months, 1 year and annually thereafter. The data are presented as cumulative deaths at each time point.
Time Frame: 30 days, 6 months, 1 year, 2 years, 3 years, 4 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 124
Participants
  30 days | 1
  6 months | 4
  1 year | 10
  2 years | 23
  3 years | 31
  4 years | 45

7. Secondary Outcome: Recurrent Heart Failure Hospitalization
Description: Recurrent heart failure hospitalization at 30 days, 6 months, 1 year and annually thereafter. The data are presented as cumulative heart failure hospitalizations at each time point.
Time Frame: 30 days , 6 months, 1 year, 2 year, 3 year, 4 year
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 124
Participants
  30 days | 3
  6 months | 10
  1 year | 15
  2 year (site-reported) | 23
  3 year (site-reported) | 29
  4 years (site-reported) | 33

8. Secondary Outcome: Reintervention Rates for Mitral Regurgitation
Description: Reintervention rates for mitral regurgitation at 30 days, 6 months, 1 year and annually thereafter. The data are presented as cumulative reintervention rates at each time point.
Time Frame: 30 days, 6 months, 1 year, 2 year, 3 year, 4 year
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 124
Participants
  30 days | 1
  6 months | 2
  1 year | 2
  2 year (site-reported) | 3
  3 year (site-reported) | 4
  4 years (site-reported) | 6

9. Secondary Outcome: Composite of Major Adverse Events (MAEs) Defined as Cardiovascular Mortality, Stroke, Myocardial Infarction, New Need for Renal Replacement Therapy, Severe Bleeding and Reintervention for Study Device Related Complications.
Description: Composite of major adverse events (MAEs) defined as cardiovascular mortality, stroke, myocardial infarction, new need for renal replacement therapy, severe bleeding and re-intervention for study device related complications at 6 months, 1 year and annually thereafter. The outcome is analyzed as the count and percentage of participants with events at each timepoint.
Time Frame: 6 months, 1 year, 2 year, 3 year, 4 year
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 124
Participants
  6 months | 16
  1 year | 23
  2 year (site-reported) | 26
  3 year (site-reported) | 33
  4 years (site-reported) | 45

10. Secondary Outcome: LVEDV by Study Visit
Description: Left ventricular end diastolic volume (LVEDV) by study visit, measured by independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline, 6 Months, 1 Year, 2 Years, 3 Years, 4 Years
Population: Participants with an LVEDV measurement available after collection of all study data for the visit.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 108
milliliters
  Baseline Visit | 181.2 (60.8)
  6-Month Visit: number analyzed (Participants) | 94
  6-Month Visit | 166.2 (61.3)
  1-Year Visit: number analyzed (Participants) | 79
  1-Year Visit | 152.8 (55.6)
  2-Year Visit: number analyzed (Participants) | 67
  2-Year Visit | 145.9 (58.5)
  3-Year Visit: number analyzed (Participants) | 54
  3-Year Visit | 151.3 (66.1)
  4-Year Visit: number analyzed (Participants) | 44
  4-Year Visit | 141.2 (63.3)

11. Secondary Outcome: Change in LVEDV, Baseline to 6-Month Visit
Description: Change in left ventricular end diastolic volume (LVEDV) from the Baseline to the 6-Month visit, measured by independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 6 Months
Population: Participants with LVEDV measurements available for both the Baseline and 6-Month visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 86
milliliters
  Baseline Visit | 187.3 (60.9)
  6-Month Visit | 169.9 (61.1)
  Change from Baseline | -17.4 (30.5)

12. Secondary Outcome: Change in LVEDV, Baseline to 1-Year Visit
Description: Change in left ventricular end diastolic volume (LVEDV) from the Baseline to the 1-Year visit, measured by independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 1 Year
Population: Participants with LVEDV measurements available for both the Baseline and 1-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 73
milliliters
  Baseline Visit | 178.0 (61.5)
  1-Year Visit | 153.3 (54.3)
  Change from Baseline | -24.6 (34.8)

13. Secondary Outcome: Change in LVEDV, Baseline to 2-Year Visit
Description: Change in left ventricular end diastolic volume (LVEDV) from the Baseline to the 2-Year visit, measured by independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 2 Years
Population: Participants with LVEDV measurements available for both the Baseline and 2-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 60
milliliters
  Baseline Visit | 182.1 (64.0)
  2-Year Visit | 153.0 (57.6)
  Change from Baseline | -29.1 (38.3)

14. Secondary Outcome: Change in LVEDV, Baseline to 3-Year Visit
Description: Change in left ventricular end diastolic volume (LVEDV) from the Baseline to the 3-Year visit, measured by independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 3 Years
Population: Participants with LVEDV measurements available for both the Baseline and 3-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 47
milliliters
  Baseline Visit | 187.6 (66.0)
  3-Year Visit | 161.5 (64.7)
  Change from Baseline | -26.1 (38.2)

15. Secondary Outcome: Change in LVEDV, Baseline to 4-Year Visit
Description: Change in left ventricular end diastolic volume (LVEDV) from the Baseline to the 4-Year visit, measured by independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 4 Years
Population: Participants with LVEDV measurements available for both the Baseline and 4-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 38
milliliters
  Baseline Visit | 174.2 (64.6)
  4-Year Visit | 147.6 (64.9)
  Change from Baseline | -26.6 (33.6)

16. Secondary Outcome: LVESV by Study Visit
Description: Left ventricular end systolic volume (LVESV) by study visit, measured by independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline, 6 Months, 1 Year, 2 Years, 3 Years, 4 Years
Population: Participants with an LVESV measurement available after collection of all study data for the visit.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 108
milliliters
  Baseline Visit | 108.7 (55.1)
  6-Month Visit: number analyzed (Participants) | 94
  6-Month Visit | 100.6 (54.0)
  1-Year Visit: number analyzed (Participants) | 79
  1-Year Visit | 91.1 (49.4)
  2-Year Visit: number analyzed (Participants) | 67
  2-Year Visit | 86.0 (51.7)
  3-Year Visit: number analyzed (Participants) | 54
  3-Year Visit | 91.9 (57.7)
  4-Year Visit: number analyzed (Participants) | 44
  4-Year Visit | 82.3 (54.9)

17. Secondary Outcome: Change in LVESV, Baseline to 6-Month Visit
Description: Change in left ventricular end systolic volume (LVESV) from the Baseline to the 6-Month visit, measured by independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 6 Months
Population: Participants with LVESV measurements available for both the Baseline and 6-Month visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 86
milliliters
  Baseline Visit | 112.6 (56.5)
  6-Month Visit | 103.2 (54.2)
  Change from Baseline | -9.3 (22.5)

18. Secondary Outcome: Change in LVESV, Baseline to 1-Year Visit
Description: Change in left ventricular end systolic volume (LVESV) from the Baseline to the 1-Year visit, measured by independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 1 Year
Population: Participants with LVESV measurements available for both the Baseline and 1-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 73
milliliters
  Baseline Visit | 104.6 (54.9)
  1-Year Visit | 90.8 (48.1)
  Change from Baseline | -13.7 (27.0)

19. Secondary Outcome: Change in LVESV, Baseline to 2-Year Visit
Description: Change in left ventricular end systolic volume (LVESV) from the Baseline to the 2-Year visit, measured by independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 2 Years
Population: Participants with LVESV measurements available for both the Baseline and 2-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 60
milliliters
  Baseline Visit | 109.6 (59.1)
  2-Year Visit | 91.6 (51.7)
  Change from Baseline | -18.0 (30.0)

20. Secondary Outcome: Change in LVESV, Baseline to 3-Year Visit
Description: Change in left ventricular end systolic volume (LVESV) from the Baseline to the 3-Year visit, measured by independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 3 Years
Population: Participants with LVESV measurements available for both the Baseline and 3-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 47
milliliters
  Baseline Visit | 114.5 (60.1)
  6-Month Visit | 100.2 (57.4)
  Change from Baseline | -14.4 (28.9)

21. Secondary Outcome: Change in LVESV, Baseline to 4-Year Visit
Description: Change in left ventricular end systolic volume (LVESV) from the Baseline to the 4-Year visit, measured by independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 4 Years
Population: Participants with LVESV measurements available for both the Baseline and 4-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 38
milliliters
  Baseline Visit | 101.7 (59.2)
  4-Year Visit | 88.1 (56.9)
  Change from Baseline | -13.6 (30.4)

22. Secondary Outcome: PASP by Study Visit
Description: Pulmonary artery systolic pressure (PASP) by study visit, measured by independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline, 6 Months, 1 Year, 2 Years, 3 Years, 4 Years
Population: Participants with a PASP measurement available after collection of all study data for the visit.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 112
millimeters of mercury (mmHg)
  Baseline Visit | 46.4 (12.6)
  6-Month Visit: number analyzed (Participants) | 92
  6-Month Visit | 39.7 (11.2)
  1-Year Visit: number analyzed (Participants) | 76
  1-Year Visit | 39.9 (11.6)
  2-Year Visit: number analyzed (Participants) | 58
  2-Year Visit | 37.2 (11.9)
  3-Year Visit: number analyzed (Participants) | 52
  3-Year Visit | 39.8 (12.2)
  4-Year Visit: number analyzed (Participants) | 40
  4-Year Visit | 39.6 (14.1)

23. Secondary Outcome: Change in PASP, Baseline to 6-Month Visit
Description: Change in pulmonary artery systolic pressure (PASP) from the Baseline to the 6-Month visit, measured by independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 6 Months
Population: Participants with PASP measurements available for both the Baseline and 6-Month visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 89
millimeters of mercury (mmHg)
  Baseline Visit | 46.0 (12.0)
  6-Month Visit | 40.2 (11.0)
  Change from Baseline | -5.8 (12.0)

24. Secondary Outcome: Change in PASP, Baseline to 1-Year Visit
Description: Change in pulmonary artery systolic pressure (PASP) from the Baseline to the 1-Year visit, measured by independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 1 Year
Population: Participants with PASP measurements available for both the Baseline and 1-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 74
millimeters of mercury (mmHg)
  Baseline Visit | 46.4 (11.9)
  1-Year Visit | 40.2 (11.5)
  Change from Baseline | -6.2 (12.9)

25. Secondary Outcome: Change in PASP, Baseline to 2-Year Visit
Description: Change in pulmonary artery systolic pressure (PASP) from the Baseline to the 2-Year visit, measured by independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 2 Years
Population: Participants with PASP measurements available for both the Baseline and 2-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 53
millimeters of mercury (mmHg)
  Baseline Visit | 45.0 (12.2)
  2-Year Visit | 38.0 (11.9)
  Change from Baseline | -6.9 (13.8)

26. Secondary Outcome: Change in PASP, Baseline to 3-Year Visit
Description: Change in pulmonary artery systolic pressure (PASP) from the Baseline to the 3-Year visit, measured by independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 3 Years
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 50
millimeters of mercury (mmHg)
  Baseline Visit | 44.2 (12.1)
  6-Month Visit | 40.4 (12.0)
  Change from Baseline | -3.8 (14.9)

27. Secondary Outcome: Change in PASP, Baseline to 4-Year Visit
Description: Change in pulmonary artery systolic pressure (PASP) from the Baseline to the 4-Year visit, measured by independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 4 Years
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 36
millimeters of mercury (mmHg)
  Baseline Visit | 43.6 (13.8)
  4-Year Visit | 40.7 (14.3)
  Change from Baseline | -2.8 (16.1)

28. Secondary Outcome: 6MWD by Study Visit
Description: Six-minute walk distance (6MWD) by study visit
Time Frame: Baseline, 6 Months and 1 Year
Population: Participants with a 6MWD measurement available after collection of all study data for the visit
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 124
meters
  Baseline Visit | 265.4 (86.6)
  6-Month Visit: number analyzed (Participants) | 104
  6-Month Visit | 290.8 (103.3)
  1-Year Visit: number analyzed (Participants) | 82
  1-Year Visit | 312.4 (104.1)

29. Secondary Outcome: Change in 6MWD, Baseline to 6-Month Visit
Description: Change in 6-minute walk distance (6MWD) from the Baseline to the 6-Month visit
Time Frame: Baseline and 6 Months
Population: Participants with 6MWD measurements available for both the Baseline and 6-Month visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 104
meters
  Baseline Visit | 273.2 (87.5)
  6-Month Visit | 290.8 (103.3)
  Change from Baseline | 17.6 (87.6)

30. Secondary Outcome: Change in 6MWD, Baseline to 1-Year Visit
Description: Change 6-minute walk distance (6MWD) from the Baseline to the 1-Year visit
Time Frame: Baseline and 1 Year
Population: Participants with 6MWD measurements available for both the Baseline and 1-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 82
meters
  Baseline Visit | 278.1 (84.5)
  1-Year Visit | 312.4 (104.1)
  Change from Baseline | 34.3 (83.6)

31. Secondary Outcome: Change in NYHA Functional Classification
Description: NYHA Functional Classification at 6 months, 1 year and annually thereafter. NYHA Classification - The stages of heart failure: Class I - No symptoms and no limitation in ordinary physical activity. Class II - Mild symptoms and slight limitation during ordinary activity. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest. Class IV - Severe limitations. Experiences symptoms even while at rest.
Time Frame: Baseline, 6 Months, 1 Year, 2 Years, 3 Years, 4 Years
Population: The outcome is reported where data are available.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 124
Participants
  Baseline: number analyzed (Participants) | 123
  Baseline: Class I | 0
  Baseline: Class II | 49
  Baseline: Class III | 68
  Baseline: Class IV | 6
  6 Months: number analyzed (Participants) | 111
  6 Months: Class I | 49
  6 Months: Class II | 52
  6 Months: Class III | 9
  6 Months: Class IV | 1
  1 Year: number analyzed (Participants) | 102
  1 Year: Class I | 44
  1 Year: Class II | 48
  1 Year: Class III | 10
  1 Year: Class IV | 0
  2 Years: number analyzed (Participants) | 82
  2 Years: Class I | 43
  2 Years: Class II | 33
  2 Years: Class III | 6
  2 Years: Class IV | 0
  3 Years: number analyzed (Participants) | 62
  3 Years: Class I | 27
  3 Years: Class II | 25
  3 Years: Class III | 9
  3 Years: Class IV | 1
  4 Years: number analyzed (Participants) | 52
  4 Years: Class I | 24
  4 Years: Class II | 22
  4 Years: Class III | 5
  4 Years: Class IV | 1

32. Secondary Outcome: KCCQ OS Score by Study Visit
Description: Kansas City Cardiomyopathy Questionnaire Overall Summary (KCCQ OS) score by study visit. The KCCQ OS score is a validated measure summarizing a patient's overall health status based on their self-assessment of heart failure symptoms, physical limitations, social limitations, and quality of life on a 23-item, self-administered questionnaire. KCCQ OS scores range from 0 to 100, with higher scores indicating better health status.
Time Frame: Baseline, 30 Days, 6 Months and 1 Year
Population: Participants with a KCCQ OS score value available after collection of all study data for the visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 124
score on a scale
  Baseline Visit | 54.6 (21.3)
  30-Day Visit: number analyzed (Participants) | 120
  30-Day Visit | 70.7 (17.8)
  6-Month Visit: number analyzed (Participants) | 111
  6-Month Visit | 71.7 (15.3)
  1-Year Visit: number analyzed (Participants) | 96
  1-Year Visit | 72.0 (16.7)

33. Secondary Outcome: Change in KCCQ OS Score, Baseline to 30-Day Visit
Description: Change in Kansas City Cardiomyopathy Questionnaire Overall Summary (KCCQ OS) Score from the Baseline to the 30-Day visit. The KCCQ OS score is a validated measure summarizing a patient's overall health status based on their self-assessment of heart failure symptoms, physical limitations, social limitations, and quality of life on a 23-item, self-administered questionnaire. KCCQ OS scores range from 0 to 100, with higher scores indicating better health status.
Time Frame: Baseline and 30 Days
Population: Participants with KCCQ OS scores available for both the Baseline and 30-Day visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 120
score on a scale
  Baseline Visit | 54.6 (21.7)
  30-Day Visit | 70.7 (17.8)
  Change from Baseline | 16.0 (18.9)

34. Secondary Outcome: Change in KCCQ OS Score, Baseline to 6-Month Visit
Description: Change in Kansas City Cardiomyopathy Overall Summary (KCCQ OS) score from the Baseline to the 6-Month visit. The KCCQ OS score is a validated measure summarizing a patient's overall health status based on their self-assessment of heart failure symptoms, physical limitations, social limitations, and quality of life on a 23-item, self-administered questionnaire. KCCQ OS scores range from 0 to 100, with higher scores indicating better health status.
Time Frame: Baseline and 6 Months
Population: Participants with KCCQ OS scores available for both the Baseline and 6-Month visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 111
score on a scale
  Baseline Visit | 56.2 (20.8)
  6-Month Visit | 71.7 (15.3)
  Change from Baseline | 15.5 (18.5)

35. Secondary Outcome: Change in KCCQ OS Score, Baseline to 1-Year Visit
Description: Change in Kansas City Cardiomyopathy Questionnaire Overall Summary (KCCQ OS) score from the Baseline to the 1-Year visit. The KCCQ OS score is a validated measure summarizing a patient's overall health status based on their self-assessment of heart failure symptoms, physical limitations, social limitations, and quality of life on a 23-item, self-administered questionnaire. KCCQ OS scores range from 0 to 100, with higher scores indicating better health status.
Time Frame: Baseline and 1 Year
Population: Participants with KCCQ OS scores available for both the Baseline and 1-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 96
score on a scale
  Baseline Visit | 56.1 (20.8)
  1-Year Visit | 72.0 (16.7)
  Change from Baseline | 15.9 (17.4)

36. Secondary Outcome: EQ5D VAS Score by Study Visit
Description: EQ5D visual analogue scale (VAS) score by study visit. The EQ5D is a validated, self-administered quality of life questionnaire including a VAS that records the respondent's self-rated health status on a graduated scale (0-100), with higher scores for higher health-related quality of life.
Time Frame: Baseline, 30 Days, 6 Months and 1 Year
Population: Participants with an EQ5D VAS score available after collection of all study data for the visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 123
score on a scale
  Baseline Visit | 62.8 (21.7)
  30-Day Visit: number analyzed (Participants) | 117
  30-Day Visit | 74.3 (19.6)
  6-Month Visit: number analyzed (Participants) | 111
  6-Month Visit | 75.1 (17.6)
  1-Year Visit: number analyzed (Participants) | 96
  1-Year Visit | 73.4 (20.3)

37. Secondary Outcome: Change in EQ5D VAS Score, Baseline to 30-Day Visit
Description: Change in EQ5D visual analogue scale (VAS) score from the Baseline to the 30-Day visit. The EQ5D is a validated, self-administered quality of life questionnaire including a VAS that records the respondent's self-rated health status on a graduated scale (0-100), with higher scores for higher health-related quality of life.
Time Frame: Baseline and 30 Days
Population: Participants with EQ5D VAS score values available for both the Baseline and 30-Day visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 116
score on a scale
  Baseline Visit | 62.4 (22.1)
  30-Day Visit | 74.2 (19.7)
  Change from Baseline | 11.8 (20.7)

38. Secondary Outcome: Change in EQ5D VAS Score, Baseline to 6-Month Visit
Description: Change in EQ5D visual analogue scale (VAS) score from the Baseline to the 6-Month visit. The EQ5D is a validated, self-administered quality of life questionnaire including a VAS that records the respondent's self-rated health status on a graduated scale (0-100), with higher scores for higher health-related quality of life.
Time Frame: Baseline and 6 Months
Population: Participants with EQ5D VAS score values available for both the Baseline and 6-Month visits after collection of all study data for these visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 110
score on a scale
  Baseline Visit | 63.9 (21.4)
  6-Month Visit | 75.3 (17.6)
  Change from Baseline | 11.5 (19.2)

39. Secondary Outcome: Change in EQ5D VAS Score, Baseline to 1-Year Visit
Description: Change in EQ5D visual analogue scale (VAS) score from the Baseline to the 1-Year visit. The EQ5D is a validated, self-administered quality of life questionnaire including a VAS that records the respondent's self-rated health status on a graduated scale (0-100), with higher scores for higher health-related quality of life.
Time Frame: Baseline and 1 Year
Population: Participants with EQ5D VAS score values available for both the Baseline and 1-Year visits after collection of all study data for these visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 95
score on a scale
  Baseline Visit | 64.2 (21.4)
  1-Year Visit | 73.4 (20.4)
  Change from Baseline | 9.2 (21.8)

40. Secondary Outcome: NT-proBNP by Study Visit
Description: N-terminal pro-B-type natriuretic peptide (NT-proBNP) level by study visit.
Time Frame: Baseline, 6 Months, 1 Year, 2 Years, 3 Years, 4 Years
Population: Participants with an NT-proBNP measurement available after collection of all study data for the visit
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/ml)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 36
picograms per milliliter (pg/ml)
  Baseline Visit | 4148.7 (6430.8)
  6-Month Visit: number analyzed (Participants) | 28
  6-Month Visit | 2835.0 (3817.8)
  1-Year Visit: number analyzed (Participants) | 33
  1-Year Visit | 2620.2 (3061.1)
  2-Year Visit: number analyzed (Participants) | 12
  2-Year Visit | 2038.2 (2636.6)
  3-Year Visit: number analyzed (Participants) | 12
  3-Year Visit | 2425.2 (2024.8)
  4-Year Visit: number analyzed (Participants) | 11
  4-Year Visit | 1837.6 (1718.0)

41. Secondary Outcome: Change in NT-proBNP, Baseline to 6-Month Visit
Description: Change in N-terminal pro-B-type natriuretic peptide (NT-proBNP) from the Baseline to the 6-Month visit
Time Frame: Baseline and 6 Months
Population: Participants with NT-proBNP measurements available for both the Baseline and 6-Month visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/ml)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 25
picograms per milliliter (pg/ml)
  Baseline Visit | 3594.7 (6145.9)
  6-Month Visit | 2695.5 (3934.3)
  Change from Baseline | -899.2 (6381.3)

42. Secondary Outcome: Change in NT-proBNP, Baseline to 1-Year Visit
Description: Change in N-terminal pro-B-type natriuretic peptide (NT-proBNP) from the Baseline to the 1-Year visit
Time Frame: Baseline and 1 Year
Population: Participants with NT-proBNP measurements available for both the Baseline and 1-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/ml)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 26
picograms per milliliter (pg/ml)
  Baseline Visit | 3450.8 (6030.8)
  1-Year Visit | 2129.2 (1820.5)
  Change from Baseline | -1321.6 (5163.6)

43. Secondary Outcome: Change in NT-proBNP, Baseline to 2-Year Visit
Description: Change in N-terminal pro-B-type natriuretic peptide (NT-proBNP) from the Baseline to the 2-Year visit
Time Frame: Baseline and 2 Years
Population: Participants with NT-proBNP measurements available for both the Baseline and 2-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/ml)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 11
picograms per milliliter (pg/ml)
  Baseline Visit | 2505.9 (2607.7)
  2-Year Visit | 1313.1 (841.0)
  Change from Baseline | -1192.8 (2186.3)

44. Secondary Outcome: Change in NT-proBNP, Baseline to 3-Year Visit
Description: Change in N-terminal pro-B-type natriuretic peptide (NT-proBNP) from the Baseline to the 3-Year visit
Time Frame: Baseline and 3 Years
Population: Participants with NT-proBNP measurements available for both the Baseline and 3-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/ml)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 10
picograms per milliliter (pg/ml)
  Baseline Visit | 2802.4 (2801.1)
  3-Year Visit | 2513.6 (2083.5)
  Change from Baseline | -288.8 (2926.2)

45. Secondary Outcome: Change in NT-proBNP, Baseline to 4-Year Visit
Description: Change in N-terminal pro-B-type natriuretic peptide (NT-proBNP) from the Baseline to the 4-Year visit
Time Frame: Baseline and 4 Years
Population: Participants with NT-proBNP measurements available for both the Baseline and 4-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/ml)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 8
picograms per milliliter (pg/ml)
  Baseline Visit | 2239.8 (2977.4)
  4-Year Visit | 1489.4 (991.4)
  Change from Baseline | -750.4 (2311.0)

46. Secondary Outcome: BNP by Study Visit
Description: Brain natriuretic peptide (BNP) level by study visit
Time Frame: Baseline, 6 Months, 1 Year, 2 Years, 3 Years, 4 Years
Population: Participants with a BNP measurement available after collection of all study data for the visit
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/ml)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 87
picograms per milliliter (pg/ml)
  Baseline Visit | 839.5 (904.4)
  6-Month Visit: number analyzed (Participants) | 79
  6-Month Visit | 588.0 (734.8)
  1-Year Visit: number analyzed (Participants) | 61
  1-Year Visit | 569.3 (923.8)
  2-Year Visit: number analyzed (Participants) | 59
  2-Year Visit | 472.4 (531.2)
  3-Year Visit: number analyzed (Participants) | 43
  3-Year Visit | 500.0 (610.3)
  4-Year Visit: number analyzed (Participants) | 34
  4-Year Visit | 451.3 (456.6)

47. Secondary Outcome: Change in BNP, Baseline to 6-Month Visit
Description: Change in brain natriuretic peptide (BNP) level from the Baseline to the 6-Month visit
Time Frame: Baseline and 6 Months
Population: Participants with BNP measurements available for both the Baseline and 6-Month visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/ml)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 75
picograms per milliliter (pg/ml)
  Baseline Visit | 813.5 (836.7)
  6-Month Visit | 606.6 (749.6)
  Change from Baseline | -206.9 (607.5)

48. Secondary Outcome: Change BNP, Baseline to 1-Year Visit
Description: Change in brain natriuretic peptide (BNP) level from the Baseline to the 1-Year visit
Time Frame: Baseline and 1 Year
Population: Participants with BNP measurements available for both the Baseline and 1-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/ml)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 58
picograms per milliliter (pg/ml)
  Baseline Visit | 746.7 (795.6)
  1-Year Visit | 585.4 (944.8)
  Change from Baseline | -161.3 (784.7)

49. Secondary Outcome: Change in BNP, Baseline to 2-Year Visit
Description: Change in brain natriuretic peptide (BNP) level from the Baseline to the 2-Year visit
Time Frame: Baseline and 2 Years
Population: Participants with BNP measurements available for both the Baseline and 2-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/ml)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 56
picograms per milliliter (pg/ml)
  Baseline Visit | 720.6 (751.3)
  2-Year Visit | 470.8 (538.6)
  Change from Baseline | -249.8 (684.4)

50. Secondary Outcome: Change in BNP, Baseline to 3-Year Visit
Description: Change in brain natriuretic peptide (BNP) level from the Baseline to the 3-Year visit
Time Frame: Baseline and 3 Years
Population: Participants with BNP measurements available for both the Baseline and 3-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/ml)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 41
picograms per milliliter (pg/ml)
  Baseline Visit | 744.2 (807.5)
  3-Year Visit | 510.4 (623.1)
  Change from Baseline | -233.9 (617.6)

51. Secondary Outcome: Change in BNP, Baseline to 4-Year Visit
Description: Change in brain natriuretic peptide (BNP) level from the Baseline to the 4-Year visit
Time Frame: Baseline and 4 Years
Population: Participants with BNP measurements available for both the Baseline and 4-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/ml)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 32
picograms per milliliter (pg/ml)
  Baseline Visit | 602.3 (588.1)
  4-Year Visit | 458.3 (468.0)
  Change from Baseline | -144.0 (572.6)

52. Secondary Outcome: Change in Tricuspid Regurgitation From Baseline
Description: Change in tricuspid regurgitation (TR) severity grade from the Baseline visit. TR severity was graded on a 5-point scale (none/trace, mild, mild-moderate, moderate-severe, severe) by independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging.
Time Frame: 6 Month, 1 Year, 2 Years, 3 Years, 4 Years
Population: Participants with TR severity grades available for both the Baseline and follow-up visit after collection of all study data for these visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 109
Participants
  6-Month Visit: 3 Grade Increase | 0
  6-Month Visit: 2 Grade Increase | 1
  6-Month Visit: 1 Grade Increase | 14
  6-Month Visit: No Change | 58
  6-Month Visit: 1 Grade Decrease | 35
  6-Month Visit: 2 Grade Decrease | 1
  6-Month Visit: 3 Grade Decrease | 0
  1-Year Visit: number analyzed (Participants) | 91
  1-Year Visit: 3 Grade Increase | 1
  1-Year Visit: 2 Grade Increase | 1
  1-Year Visit: 1 Grade Increase | 8
  1-Year Visit: No Change | 49
  1-Year Visit: 1 Grade Decrease | 30
  1-Year Visit: 2 Grade Decrease | 2
  1-Year Visit: 3 Grade Decrease | 0
  2-Year Visit: number analyzed (Participants) | 70
  2-Year Visit: 3 Grade Increase | 1
  2-Year Visit: 2 Grade Increase | 1
  2-Year Visit: 1 Grade Increase | 8
  2-Year Visit: No Change | 40
  2-Year Visit: 1 Grade Decrease | 18
  2-Year Visit: 2 Grade Decrease | 2
  2-Year Visit: 3 Grade Decrease | 0
  3-Year Visit: number analyzed (Participants) | 59
  3-Year Visit: 3 Grade Increase | 1
  3-Year Visit: 2 Grade Increase | 4
  3-Year Visit: 1 Grade Increase | 7
  3-Year Visit: No Change | 34
  3-Year Visit: 1 Grade Decrease | 12
  3-Year Visit: 2 Grade Decrease | 1
  3-Year Visit: 3 Grade Decrease | 0
  4-Year Visit: number analyzed (Participants) | 46
  4-Year Visit: 3 Grade Increase | 1
  4-Year Visit: 2 Grade Increase | 3
  4-Year Visit: 1 Grade Increase | 4
  4-Year Visit: No Change | 27
  4-Year Visit: 1 Grade Decrease | 10
  4-Year Visit: 2 Grade Decrease | 1
  4-Year Visit: 3 Grade Decrease | 0

53. Secondary Outcome: Mitral EROA by Study Visit
Description: Mitral effective regurgitant orifice area (EROA) by study visit, measured using the proximal isovelocity surface area (PISA) method during independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline, 30 Days, 6 Months, 1 Year, 2 Years, 3 Years, 4 Years
Population: Participants with a mitral EROA measurement available after collection of all study data for the visit
Measure: Mean (Standard Deviation); unit: square centimeters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 101
square centimeters
  Baseline Visit | 0.38 (0.15)
  30-Day Visit: number analyzed (Participants) | 25
  30-Day Visit | 0.17 (0.21)
  6-Month Visit: number analyzed (Participants) | 19
  6-Month Visit | 0.15 (0.06)
  1-Year Visit: number analyzed (Participants) | 10
  1-Year Visit | 0.18 (0.06)
  2-Year Visit: number analyzed (Participants) | 6
  2-Year Visit | 0.19 (0.03)
  3-Year Visit: number analyzed (Participants) | 6
  3-Year Visit | 0.24 (0.13)
  4-Year Visit: number analyzed (Participants) | 5
  4-Year Visit | 0.25 (0.10)

54. Secondary Outcome: Change in Mitral EROA, Baseline to 30-Day Visit
Description: Change in mitral effective regurgitant orifice area (EROA) from the Baseline to the 30-Day visit, measured using the proximal isovelocity surface area (PISA) method during independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 30 Days
Population: Participants with mitral EROA measurements available for both the Baseline and 30-Day visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: square centimeters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 24
square centimeters
  Baseline Visit | 0.40 (0.17)
  30-Day Visit | 0.17 (0.21)
  Change from Baseline | -0.24 (0.22)

55. Secondary Outcome: Change in Mitral EROA, Baseline to 6-Month Visit
Description: Change in mitral effective regurgitant orifice area (EROA) from the Baseline to the 6-Month visit, measured using the proximal isovelocity surface area (PISA) method during independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 6 Months
Population: Participants with mitral EROA measurements available for both the Baseline and 6-Month visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: square centimeters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 15
square centimeters
  Baseline Visit | 0.40 (0.15)
  6-Month Visit | 0.14 (0.06)
  Change from Baseline | -0.27 (0.15)

56. Secondary Outcome: Change in Mitral EROA, Baseline to 1-Year Visit
Description: Change in mitral effective regurgitant orifice area (EROA) from the Baseline to the 1-Year visit, , measured using the proximal isovelocity surface area (PISA) method during independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 1 Year
Population: Participants with mitral EROA measurements available for both the Baseline and 1-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: square centimeters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 9
square centimeters
  Baseline Visit | 0.41 (0.21)
  1-Year Visit | 0.18 (0.06)
  Change from Baseline | -0.22 (0.20)

57. Secondary Outcome: Change in Mitral EROA, Baseline to 2-Year Visit
Description: Change in mitral effective regurgitant orifice area (EROA) from the Baseline to the 2-Year visit, measured using the proximal isovelocity surface area (PISA) method during independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 2 Years
Population: Participants with mitral EROA measurements available for both the Baseline and 2-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: square centimeters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 6
square centimeters
  Baseline Visit | 0.35 (0.08)
  2-Year Visit | 0.19 (0.03)
  Change from Baseline | -0.16 (0.06)

58. Secondary Outcome: Change in Mitral EROA, Baseline to 3-Year Visit
Description: Change in mitral effective regurgitant orifice area (EROA) from the Baseline to the 3-Year visit, measured using the proximal isovelocity surface area (PISA) method during independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 3 Years
Population: Participants with mitral EROA measurements available for both the Baseline and 3-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: square centimeters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 5
square centimeters
  Baseline Visit | 0.36 (0.04)
  3-Year Visit | 0.25 (0.14)
  Change from Baseline | -0.11 (0.14)

59. Secondary Outcome: Change in Mitral EROA, Baseline to 4-Year Visit
Description: Change in mitral effective regurgitant orifice area (EROA) from the Baseline to the 4-Year visit, measured using the proximal isovelocity surface area (PISA) method during independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 4 Years
Population: Participants with mitral EROA measurements available for both the Baseline and 4-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: square centimeters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 4
square centimeters
  Baseline Visit | 0.44 (0.08)
  4-Year Visit | 0.28 (0.09)
  Change from Baseline | -0.16 (0.02)

60. Secondary Outcome: Mitral Regurgitant Volume by Study Visit
Description: Mitral regurgitant volume by study visit, measured using the proximal isovelocity surface area (PISA) method during independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline, 30 Days, 6 Months, 1 Year, 2 Years, 3 Years, 4 Years
Population: Participants with a mitral regurgitant volume measurement available after collection of all study data for the visit
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 99
milliliters
  Baseline Visit | 57.3 (19.7)
  30-Day Visit: number analyzed (Participants) | 25
  30-Day Visit | 25.2 (18.7)
  6-Month Visit: number analyzed (Participants) | 19
  6-Month Visit | 25.3 (11.2)
  1-Year Visit: number analyzed (Participants) | 10
  1-Year Visit | 30.1 (10.1)
  2-Year Visit: number analyzed (Participants) | 6
  2-Year Visit | 31.0 (7.3)
  3-Year Visit: number analyzed (Participants) | 6
  3-Year Visit | 38.0 (18.8)
  4-Year Visit: number analyzed (Participants) | 5
  4-Year Visit | 37.8 (16.7)

61. Secondary Outcome: Change in Mitral Regurgitant Volume, Baseline to 30-Day Visit
Description: Change in mitral regurgitant volume from the Baseline to the 30-Day visit, measured using the proximal isovelocity surface area (PISA) method during independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 30 Days
Population: Participants with mitral regurgitant volume measurements available for both the Baseline and 30-Day visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 23
milliliters
  Baseline Visit | 62.5 (18.3)
  30-Day Visit | 24.3 (19.3)
  Change from Baseline | -38.2 (23.8)

62. Secondary Outcome: Change in Mitral Regurgitant Volume, Baseline to 6-Month Visit
Description: Change in mitral regurgitant volume from the Baseline to the 6-Month visit, measured using the proximal isovelocity surface area (PISA) method during independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 6 Months
Population: Participants with mitral regurgitant volume measurements available for both the Baseline and 6-Month visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 15
milliliters
  Baseline Visit | 62.8 (16.4)
  6-Month Visit | 22.8 (10.2)
  Change from Baseline | -40.0 (19.5)

63. Secondary Outcome: Change in Mitral Regurgitant Volume, Baseline to 1-Year Visit
Description: Change in mitral regurgitant volume from the Baseline to the 1-Year visit, measured using the proximal isovelocity surface area (PISA) method during independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 1 Year
Population: Participants with mitral regurgitant volume measurements available for both the Baseline and 1-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 9
milliliters
  Baseline Visit | 61.5 (16.0)
  1-Year Visit | 30.3 (10.7)
  Change from Baseline | -31.2 (17.6)

64. Secondary Outcome: Change in Mitral Regurgitant Volume, Baseline to 2-Year Visit
Description: Change in mitral regurgitant volume from the Baseline to the 2-Year visit, measured using the proximal isovelocity surface area (PISA) method during independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 2 Years
Population: Participants with mitral regurgitant volume measurements available for both the Baseline and 2-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 6
milliliters
  Baseline Visit | 54.6 (17.2)
  2-Year Visit | 31.0 (7.3)
  Change from Baseline | -23.5 (14.4)

65. Secondary Outcome: Change in Mitral Regurgitant Volume, Baseline to 3-Year Visit
Description: Change in mitral regurgitant volume from the Baseline to the 3-Year visit, measured using the proximal isovelocity surface area (PISA) method during independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 3 Years
Population: Participants with mitral regurgitant volume measurements available for both the Baseline and 3-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 5
milliliters
  Baseline Visit | 59.9 (13.5)
  3-Year Visit | 40.1 (20.2)
  Change from Baseline | -19.8 (17.1)

66. Secondary Outcome: Change in Mitral Regurgitant Volume, Baseline to 4-Year Visit
Description: Change in mitral regurgitant volume from the Baseline to the 4-Year visit, measured using the proximal isovelocity surface area (PISA) method during independent echocardiographic core lab review of transthoracic echocardiography (TTE) imaging
Time Frame: Baseline and 4 Years
Population: Participants with mitral regurgitant volume measurements available for both the Baseline and 4-Year visits after collection of all study data for these visits
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
Number analyzed (Participants) | 4
milliliters
  Baseline Visit | 74.2 (9.0)
  4-Year Visit | 41.7 (16.5)
  Change from Baseline | -32.5 (11.4)

ADVERSE EVENTS:
Time Frame: 4 year follow up
Description: All adverse events, including all-cause mortality, are reported through the exact 4-year day (day 1460)
Arm/Group | Edwards PASCAL Transcatheter Mitral Valve Repair System
All-Cause Mortality (participants affected / at risk) | 45/124
Serious Adverse Events (participants affected / at risk) | 94/124
Other Adverse Events (participants affected / at risk) | 33/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edwards PASCAL Transcatheter Mitral Valve Repair System (N=124)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 13 (16)
Acute left ventricular failure (Cardiac disorders) | 3 (3)
Angina pectoris (Cardiac disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 12 (13)
Bacteraemia (Infections and infestations) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Blood glucose increased (Investigations) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
COVID-19 (Infections and infestations) | 5 (5)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1)
Gallstone ileus (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 11 (14)
Haemorrhage (Vascular disorders) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Post stroke epilepsy (Nervous system disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 9 (11)
Chest pain (General disorders) | 4 (4)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Dementia (Nervous system disorders) | 1 (1)
Device dislocation (Product Issues) | 4 (4)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1)
Pharyngeal injury (Injury, poisoning and procedural complications) | 1 (1)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1)
Cardiac arrest (Cardiac disorders) | 7 (8)
Cardiorenal syndrome (Cardiac disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Heart transplant (Surgical and medical procedures) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (3)
Atrial thrombosis (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 2 (2)
Death (General disorders) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Middle cerebral artery stroke (Nervous system disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 7 (8)
Multiple organ dysfunction syndrome (General disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 8 (8)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 10 (10)
Cardiac failure congestive (Cardiac disorders) | 8 (9)
Chronic left ventricular failure (Cardiac disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 8 (10)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Mitral valve stenosis (Cardiac disorders) | 1 (1)
Pelvic haematoma (Reproductive system and breast disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
Pharyngeal haematoma (Injury, poisoning and procedural complications) | 1 (1)
Pleomorphic liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 3 (3)
Poor peripheral circulation (Vascular disorders) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Asthenia (General disorders) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
Arthritis infective (Infections and infestations) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 2 (2)
Haematoma (Vascular disorders) | 2 (2)
International normalised ratio increased (Investigations) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 3 (3)
Cardiogenic shock (Cardiac disorders) | 4 (4)
Gastritis (Gastrointestinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Nosocomial infection (Infections and infestations) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 3 (3)
Abscess limb (Infections and infestations) | 1 (1)
Device related thrombosis (General disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Arrhythmic storm (Cardiac disorders) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 4 (4)
Cardiac failure (Cardiac disorders) | 18 (43)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Device embolisation (General disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2)
Seizure (Nervous system disorders) | 1 (1)
Renal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 6 (6)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 4 (4)
Respiratory tract infection (Infections and infestations) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (4)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (5)
Septic shock (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 6 (7)
Viral infection (Infections and infestations) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1)
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 (1)
Urethral injury (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Transplant evaluation (Investigations) | 1 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Syncope (Nervous system disorders) | 1 (2)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 4 (4)
Shock (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edwards PASCAL Transcatheter Mitral Valve Repair System (N=124)
Atrial fibrillation (Cardiac disorders) | 11 (13)
Cardiac failure (Cardiac disorders) | 10 (10)
Urinary tract infection (Infections and infestations) | 9 (11)
Acute kidney injury (Renal and urinary disorders) | 7 (7)
Hypotension (Vascular disorders) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT03170349/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT03170349/SAP_001.pdf